CLINICAL TRIAL: NCT02414035
Title: A Monitor System for the Safety of Dabigatran Anticoagulation Treatment in Nonvalvular Atrial Fibrillation
Brief Title: Monitor System for the Safety of Dabigatran Treatment
Acronym: MISSION-AF
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2014ZX09303305
Record Dates: First submitted 2015-03-25; First posted 2015-04-10 (Estimated); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; anticoagulation; Dabigatran
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples with DNA for genetic variants test which could contribute to interindividual variability in blood concentrations of the active metabolite of dabigatran etexilate and influence the safety and efficacy of dabigatran.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine whether dabigatran is associated with higher risk of bleeding in Asia area especially in China clinical practice and whether it need to set up a monitor system.

DETAILED DESCRIPTION:
Dabigatran is administered in a fixed does without laboratory monitoring and is being compared with warfarin (international normalized ratio, but only hundreds of evidence from Asia events in several multicenter, prospective, randomized trails. It remains unclear that whether Dabigatran is safety in China clinical practice and no need of monitor test. We identified participants as those diagnosed as having nonvalved atrial fibrillation, and who initiated dabigatran after diagnosis.We followed up each individual from the first prescription of dabigatran until discontinued use or switch of anticoagulants, death, or other outcomes or until one year later. We categorized bleeding events as major and minor events according to anatomical position. We defined time to bleeding as days between the first dabigatran prescription and the date of the bleeding event. We analyzed the time to the first bleeding event, as well as the time to the first major hemorrhage, intracranial hemorrhage, gastrointestinal bleeding, hematuria, vaginal bleeding, hemarthrosis, hemoptysis, and epistaxis.

ELIGIBILITY:
Inclusion Criteria:

1. Age>18 y at entry
2. AF documented as follows: The patients has a symptomatic episode of paroxysmal or persistent AF documented by 12-lead ECG, rhythm strip, pacemaker/implantable cardioverter-defibrillator electrogram, or Holter ECG
3. In addition to documented AF, patients must have ≥1 CHADS2-VAS scores
4. We identified participants as those diagnosed as having AF, and who initiated dabigatran after diagnosis
5. Written, informed consent

Exclusion Criteria:

1. History of heart valve disorders (ie, prosthetic valve or hemodynamically relevant valve disease)
2. Severe, disabling stroke, or any stroke within the previous 14d
3. Acute coronary syndrome within 1 year in AF patients
4. Conditions associated with an increased risk of bleeding

   1. Major surgery in the previous month
   2. History of intracranial, intraocular, spinal, retroperitoneal or atraumatic intra-articular bleeding
   3. Gastrointestinal hemorrhage or hematuria
5. Severe renal impairment (estimated creatinine clearace≤30ml/min)
6. Severe liver dysfunction
7. Alcohol abuse or drug addiction
8. Patients who have received an investigational drug at this time
9. Patients considered unreliable by the investigator or have a life expectancy less than the expected duration of the trail

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We identified participants as those diagnosed as having artrial fibrillation, and who initiated dabigatran after diagnosis. The diagnosis of AF was defined as having inpatient or outpatient claims with primary or secondary International Classification of Diseases, Ninth Revision(ICD-9), code427.31.12. The CHADS2-VAS score is calculated as the sum of all points for a given patient and need >=1. A history of previous stroke or transient ischemic attack is assigned 2 points; congestive heart failure, hypertension, age of 75 years or older, and diabetes are each assigned 1 point.
Sampling Method: Non-Probability Sample
Enrollment: 1496 (Actual)
Dates: Start 2015-03-22 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-04-18 (Actual)

PRIMARY OUTCOMES:
Major bleeding events | up to 12 months (or) years
  Any of the following events happened: intracranial hemorrhage, hemoperitoneum, and inpatient or emergency department stays for gastrointestinal, hematuria,or NOS hemorrhage
Minor bleeding events | up to 12 months (or) years
  Any of the following events happened: epistaxis, hemoptysis, vaginal hemorrhage, hemarthrosis and any outpatient claim for hematuria, gastrointestinal, and NOS hemorrhage.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao s Cheng, MD,PhD, Principal Investigator — The second hospital affillated of Nanchang University
Locations (1):
- The second hospital affillated of Nanchang University, Nanchang, Jiangxi, China

REFERENCES:
- [Background] Oldgren J, Healey JS, Ezekowitz M, Commerford P, Avezum A, Pais P, Zhu J, Jansky P, Sigamani A, Morillo CA, Liu L, Damasceno A, Grinvalds A, Nakamya J, Reilly PA, Keltai K, Van Gelder IC, Yusufali AH, Watanabe E, Wallentin L, Connolly SJ, Yusuf S; RE-LY Atrial Fibrillation Registry Investigators. Variations in cause and management of atrial fibrillation in a prospective registry of 15,400 emergency department patients in 46 countries: the RE-LY Atrial Fibrillation Registry. Circulation. 2014 Apr 15;129(15):1568-76. doi: 10.1161/CIRCULATIONAHA.113.005451. Epub 2014 Jan 24. PMID 24463370
- [Background] Steinberg BA, Piccini JP. Anticoagulation in atrial fibrillation. BMJ. 2014 Apr 14;348:g2116. doi: 10.1136/bmj.g2116. PMID 24733535
- [Background] Ezekowitz MD, Connolly S, Parekh A, Reilly PA, Varrone J, Wang S, Oldgren J, Themeles E, Wallentin L, Yusuf S. Rationale and design of RE-LY: randomized evaluation of long-term anticoagulant therapy, warfarin, compared with dabigatran. Am Heart J. 2009 May;157(5):805-10, 810.e1-2. doi: 10.1016/j.ahj.2009.02.005. PMID 19376304
- [Background] Reilly PA, Lehr T, Haertter S, Connolly SJ, Yusuf S, Eikelboom JW, Ezekowitz MD, Nehmiz G, Wang S, Wallentin L; RE-LY Investigators. The effect of dabigatran plasma concentrations and patient characteristics on the frequency of ischemic stroke and major bleeding in atrial fibrillation patients: the RE-LY Trial (Randomized Evaluation of Long-Term Anticoagulation Therapy). J Am Coll Cardiol. 2014 Feb 4;63(4):321-8. doi: 10.1016/j.jacc.2013.07.104. Epub 2013 Sep 27. PMID 24076487
- [Background] Graham DJ, Reichman ME, Wernecke M, Zhang R, Southworth MR, Levenson M, Sheu TC, Mott K, Goulding MR, Houstoun M, MaCurdy TE, Worrall C, Kelman JA. Cardiovascular, bleeding, and mortality risks in elderly Medicare patients treated with dabigatran or warfarin for nonvalvular atrial fibrillation. Circulation. 2015 Jan 13;131(2):157-64. doi: 10.1161/CIRCULATIONAHA.114.012061. Epub 2014 Oct 30. PMID 25359164
- [Derived] Zhou W, Wang T, Zhu LJ, Wen MH, Hu LH, Huang X, You CJ, Li JX, Wu YQ, Wu QH, Bao HH, Cheng XS. Peripheral leukocyte count and risk of bleeding in patients with non-valvular atrial fibrillation taking dabigatran: a real-world study. Chin Med J (Engl). 2019 Sep 20;132(18):2150-2156. doi: 10.1097/CM9.0000000000000423. PMID 31490268